CLINICAL TRIAL: NCT04009148
Title: Cascade Testing in Families With Newly Diagnosed Hereditary Breast and Ovarian Cancer Syndrome
Status: Active, not recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 17-01135
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: BRCA-Mutated Ovarian Carcinoma; BRIP1 Gene Mutation; MSH2 A636P; MLH1 Gene Mutation; MSH6 Gene Mutation; PMS2 Gene Mutation; EPCAM; RAD51C Gene Mutation

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: None Retained — Living carriers of pathogenic mutations associated with HBOC and LS, and their blood relatives (first- and second-degree, and first cousins)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Successful Cascade Testing: Genetic counselor contacts relatives and offers participation in study. Relative accepts and genetic testing in performed.
  Interventions: Other: CASCADE genetic screening
- Relative Declines Genetic Testing: Genetic counselor contacts relatives and offers participation in study. Relative declines and genetic testing is not performed.
  Interventions: Other: CASCADE genetic screening

INTERVENTIONS:
Other: CASCADE genetic screening — Family-based cohort of mutation carriers, blood relatives who test negative, and untested blood relatives

SUMMARY:
Identification of BRCA mutations in ovarian cancer patients may help guide cancer therapies, prognosis, post-operative screening, and other preventative treatments beyond the initial diagnosis. Likewise, genetic testing of ovarian cancer patients for these germline mutations provides invaluable information for families regarding cancer risk, genetic testing, and subsequently indication for risk-reducing surgery. Cascade testing provides a unique opportunity to identify carriers of a deleterious BRCA mutation which can allow for surgical and chemoprevention of prevention of ovarian cancer. There is currently no literature on the rates of referral for the family members.

DETAILED DESCRIPTION:
The objective of this study is to perform a pilot study, offering referral to a genetic counseling and genetic testing for family members of a probands known to have a mutation in BRCA1 or BRCA2. In addition to BRCA1 and BRCA2, the NCCN suggests consideration of risk-reducing surgery for mutations in BRIP1, MSH2, MLH1, MSH6, PMS2, EPCAM, RAD51C, RAD51D, investigators will include these subjects as well in the study.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must have a diagnosis of epithelial ovarian cancer, Fallopian tube caner or primary peritoneal cancer with a known pathogenic genetic mutation.
* All subjects must agree to participate.
* All subjects must have first or second degree relatives who have not been diagnosed with the same genetic mutation.
* A previous diagnosis of cancer in the subject's first or second degree relative is allowed.

Exclusion Criteria:

* Subjects whose first and/or second degree relatives have already been tested with the subject's known mutations, and no other viable family members are available for testing.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: First or second degree faamily member with any of the following mutations: BRCA mutation, SH6, PMS2, EPCAM, RAD51C, RAD51D mutations
Sampling Method: Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2027-04-23 (Estimated)

PRIMARY OUTCOMES:
Establishing the CASCADE Cohort | 1 Year
  Number of relatives with successful cascade testing

CONTACTS AND LOCATIONS:
Overall Officials: Bhavana Pothuri, MD, Principal Investigator — New York Langone Medical Center
Locations (1):
- NYU Langone Health, New York, New York, United States